CLINICAL TRIAL: NCT01020656
Title: Maintenance of Anticoagulant and Antiplatelet Agents for Patients Undergoing Vitreoretinal Surgery
Brief Title: Anticoagulant and Antiplatelet Agents in Patients Undergoing Vitreoretinal Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Professor Catherine Creuzot-Garcher, Centre Hospitalier Universitaire Dijon
Other Study IDs: MARIE02
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Retinal Detachment
Keywords: anticoagulant agents; antiplatelet agents; vitreoretinal surgery; Patients suffered from retinal detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- group 1: patients with no anticoagulants used as the control group
- group 2: patients treated with anticoagulant therapy (warfarin, fluindone, acenocoumarol)
- group 3: patients treated with aspirin
- group 4: patients treated with clopidogrel therapy
- group 5: patients treated with both anticoagulant and aspirin medications
- group 6: patients treated with both anticoagulant and clopidogrel medications
- group 7: patients treated with both aspirin and clopidogrel medications

SUMMARY:
Purpose: To establish the prevalence of anticoagulant, aspirin, and clopidogrel use in patients undergoing vitreoretinal surgery, and to compare the outcome of peribulbar anesthesia between users and non-users.

ELIGIBILITY:
Inclusion Criteria:

* Take or no anticoagulant treatment before surgery,
* Vitreoretinal surgery

Exclusion Criteria:none

* No surgery
* Anesthetic complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We analyzed the chart of 239 eyes (206 patients) which underwent posterior segment surgery with peribulbar anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Unit CHU Dijon, Dijon, Burgundy, France